CLINICAL TRIAL: NCT05556174
Title: Intraoperative Lung Protective Ventilation With or Without Periodic Lung Recruitment Maneuvers on Pulmonary Complications After Major Abdominal Surgery: a Prospective Randomized Controlled Study
Brief Title: Intraoperative Lung Protective Ventilation Needs Periodic Lung Recruitment Maneuvers
Acronym: REMAIN-1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2022ZSLYEC-398
Record Dates: First submitted 2022-09-14; First posted 2022-09-27 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2024-11

CONDITIONS: Postoperative Complications; Abdominal Surgery; Intraoperative Mechanical Ventilation
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intensive intraoperative lung-protective ventilation (Experimental): intraoperative lung-protective ventilation with periodic lung recruitment maneuvers
  Interventions: Other: periodic lung recruitment maneuvers
- Moderate intraoperative lung-protective ventilation (No Intervention): intraoperative lung-protective ventilation without periodic lung recruitment maneuvers

INTERVENTIONS:
Other: periodic lung recruitment maneuvers — lung recruitment maneuvers repeated every 30 minutes
  Arms: Intensive intraoperative lung-protective ventilation

SUMMARY:
Postoperative Pulmonary Complications (PPC) are common. It severely affects postoperative recovery, particularly in abdominal surgery. Several studies showed that intraoperative lung-protective ventilation with periodic lung recruitment maneuvers could reduce postoperative pulmonary complications. Other studies showed that intraoperative lung protective ventilation without periodic lung recruitment maneuvers could also reduce postoperative pulmonary complications. The purpose of this study was to compare the effects of the above two regimens on postoperative pulmonary complications.

ELIGIBILITY:
Inclusion Criteria:

1. Undergoing elective major abdominal surgery (expected duration of mechanical ventilation ≥2 h)
2. had an intermediate to high risk of developing postoperative pulmonary complications as indicated by an Assess Respiratory Risk in Surgical Patients in Catalonia score (≥26)
3. Pulse oxygen saturation in room air ≥ 94%

Exclusion Criteria:

1. younger than 18 years
2. had received invasive mechanical ventilation for longer than 1 h within the last 2 weeks prior to surgery
3. had a history of pneumonia within 1 month prior to surgery
4. had severe chronic obstructive pulmonary disease or pulmonary bullae
5. had a progressive neuromuscular illness
6. severe heart dysfunction (New York Heart Association classification ≥4)
7. with an American Society of Anesthesiologists (ASA) physical status of IV or higher
8. Intracranial hypertension
9. were pregnant (excluded by laboratory analysis)
10. were involved in other interventional studies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1060 (Actual)
Dates: Start 2022-10-09 (Actual); Primary Completion 2024-09-11 (Actual); Study Completion 2024-11-11 (Actual)

PRIMARY OUTCOMES:
Rate of respiratory failure | Day 0 to 7 after surgery
  Respiratory failure: postoperative arterial partial pressure of oxygen (PaO2) < 8 kPa (60 mmHg) on room air, a PaO2: Inhaled oxygen concentration (FI02) ratio < 40 kPa (300 mmHg) or arterial oxyhaemoglobin saturation measured with pulse oximetry < 90% and requiring oxygen therapy

SECONDARY OUTCOMES:
Rate of mild respiratory failure | Day 0 to 7 after surgery
  Mild respiratory failure: PaO2 < 60 mmHg or pulse oxygen saturation (SpO2) < 90% on room air, but SpO2 can be raised to more than 90% when inhaling oxygen through nasal catheter less than 3 L/min.
Rate of moderate respiratory failure | Day 0 to 7 after surgery
  Moderate respiratory failure: PaO2 < 60 mmHg or SpO2 < 90% when inhaling oxygen through nasal catheter less than 3 L/min, but SpO2 can be raised to more than 90% when inhaling oxygen more than 3 L/min.
Rate of severe respiratory failure | Day 0 to 7 after surgery
  Severe respiratory failure: experienced an invasive or noninvasive ventilator therapy, or PaO2 < 60 mmHg or SpO2 < 90% when administering oxygen via a nasal catheter at 3 L/min or more.
Rate of sustained hypoxaemia | Day 0 to 7 after surgery
  Sustained hypoxaemia: during a follow-up visit when the patient was awake and breathing room air, SpO2 ≤ 92% or the change of SpO2 (ΔSpO2, preoperative SpO2 minus postoperative SpO2) ≥ 5% on any three consecutive days.
Rate of modified respiratory failure | Day 0 to 7 after surgery
  Modified respiratory failure: met the criterion of moderate or severe respiratory failure, or mild respiratory failure in twice follow-up, or mild respiratory failure with sustained hypoxemia.
Rate of respiratory infections | Day 0 to 7 after surgery
  Respiratory infections: receiving antibiotics for a suspected respiratory infection and met at least one of the following criteria: new or changed sputum, new or changed lung opacities, fever, leukocyte count >12 × 109 /L
Rate of pneumonia | Day 0 to 7 after surgery
  Pneumonia: United States Centers for Disease Control definition of pneumonia
Rate of aspiration pneumonitis | Day 0 to 7 after surgery
  Aspiration pneumonitis: acute lung injury after the inhalation of regurgitated gastric contents.
Rate of pneumothorax | Intraoperative or day 0 to 7 after surgery
  Pneumothorax: air in the pleural space with no vascular bed surrounding the visceral pleura
Rate of pleural effusion | Day 0 to 7 after surgery
  Pleural effusion: chest radiograph demonstrating blunting of the costophrenic angle, loss of sharp silhouette of the ipsilateral hemidiaphragm in upright position, evidence of displacement of adjacent anatomical structures or (in supine position) a hazy opacity in one hemithorax with preserved vascular shadows
Rate of Acute Respiratory Distress Syndrome | Day 0 to 7 after surgery
  Acute Respiratory Distress Syndrome: The Berlin definition of Respiratory Distress Syndrome
Rate of Quick Sequential Organ Failure Assessment (qSOFA) ≥ 2 | Day 0 to 7 after surgery
  qSOFA ≥ 2: Two or more of: Respiratory rate ≥22/min, Altered mentation, Systolic blood pressure ≤ 100 mm Hg
Rate of Systemic Inflammatory Response Syndrome (SIRS) | Day 0 to 7 after surgery
  SIRS: Two or more of: Temperature >38°C or <36°C, Heart rate > 90/min, Respiratory rate >20/min or PaCO2<32 mmHg (4.3kPa), White blood cell count >12 000/mm3 or 10% immature bands
Rate of Major Adverse Cardiac and Cerebrovascular Events (MACCE) | Day 0 to 7 after surgery
  MACCE: Stroke, coma, non-fatal cardiac arrest, acute myocardial infarction, congestive heart failure.
Postoperative hospitalization days | Day 0 to 30 after surgery
  The duration between the operation date and the actual discharge date, days
Rate of Unexpected admission to intensive care unit (ICU) | Day 0 to 30 after surgery
  Unexpected admission to ICU: It does not include patients who enter ICU at the request of surgeons but have normal spontaneous breathing, stable circulation and no disturbance of consciousness.
Rate of death | Day 0 to 30 after surgery
  Death from any cause
Rate of intraoperative hypotension | Intraoperative, period of mechanical ventilation
  Intraoperative hypotension: mean arterial pressure (MAP) < 60 mmHg lasting more than 3 minutes
Rate of intraoperative needing for vasoconstrictor | Intraoperative, period of mechanical ventilation
  Intraoperative vasoconstrictor needs: MAP < 60 mmHg and using any catecholamines
Rate of intraoperative hypoxemia | Intraoperative, period of mechanical ventilation
  Intraoperative hypoxemia: SpO2 ≤ 92% lasting more than 3 minutes
Rate of Intraoperative bradycardia | Intraoperative, period of mechanical ventilation
  Intraoperative bradycardia: heart rate ≤ 50 bpm and the decrease of heart rate from the basic value ≥ 20% lasting more than 3 minutes
Rate of post-anesthesia care unit respiratory failure | Postoperative, during postanesthesia care unit
  Post-anesthesia care unit respiratory failure: PaO2 < 8 kPa (60 mmHg) on room air, a PaO2:FI02 ratio < 40 kPa (300 mmHg) or arterial oxyhaemoglobin saturation measured with pulse oximetry < 90% and requiring oxygen therapy
Intraoperative mechanical power | Intraoperative: after half an hour of mechanical ventilation, before the end of mechanical ventilation
  Mechanical power, J/min
PaO2 / FI02 | Intraoperative: after half an hour of mechanical ventilation, before the end of mechanical ventilation
  PaO2 / FI02, mmHg
Postoperative pulmonary complications score | Day 0 to 7 after surgery
  Postoperative pulmonary complications score: graded on a scale from 0 (no pulmonary complications) to 4 (the most severe complications).

OTHER OUTCOMES:
Dead space rate | Intraoperative: after half an hour of mechanical ventilation, before the end of mechanical ventilation
  Dead space rate (%)

CONTACTS AND LOCATIONS:
Overall Officials: Hong Li, MD, Principal Investigator — The Sixth Affiliated Hospital, Sun Yat-sen University
Locations (1):
- The Sixth Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhang NR, Zhang LZ, Chen Y, Zhang S, Li S, Gu XK, Li J, Li H. Intraoperative protective ventilation with or without periodic lung recruitment manoeuvres on pulmonary complications after major abdominal surgery (REMAIN-1): protocol for a randomised controlled trial. BMJ Open. 2025 Mar 13;15(3):e093360. doi: 10.1136/bmjopen-2024-093360. PMID 40082005